CLINICAL TRIAL: NCT02646280
Title: The Myofascial Massage in the Treatment of Chronic Non-specific Low Back Pain: the Experience of Contact
Brief Title: Myofascial Massage in the Treatment of Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Medical Director, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3791/2015
Record Dates: First submitted 2016-01-03; First posted 2016-01-05 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Low Back Pain
Keywords: Low back pain; interoceptive awareness; motor imagery; massage
MeSH Terms: conditions — Low Back Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Massage therapy and contact experience (Experimental): Traditional massage therapy consisting of different phases: surface touch, deep touch, static pressures, dynamic pressures and kneading associated with a preparation to the contact phase of the massage using the typical elements of neurocognitive rehabilitation such as motor imagery, dynamic state during which a person mentally simulates an action, and language, necessary to understand the way of perceiving and organizing sensory, cognitive and phenomenological informations by the patients and so to interpretate pain in a more articulate way.
  Interventions: Other: Massage therapy; Other: Neurocognitive rehabilitation
- Massage therapy (Active Comparator): Traditional massage therapy consisting of different phases: surface touch, deep touch, static pressures, dynamic pressures and kneading.
  Interventions: Other: Massage therapy

INTERVENTIONS:
Other: Massage therapy — Massage therapy as a treatment option to induce a relaxation and a reduction of pain and stress in patients affected by chronic low back pain.
Other: Neurocognitive rehabilitation — Provided through the association of motor imagery and the words of the physiotherapist with the aim of increasing the effectiveness of massage in reducing pain.
  Arms: Massage therapy and contact experience

SUMMARY:
The purpose of the study is to determine the effectiveness of an approach that combines massage therapy with elements of neurocognitive rehabilitation such as motor imagery and the words of the physiotherapist compared to a traditional massage therapy in reducing pain in patients with chronic low back pain (CLBP) and to evaluate if and how the pain reduction is linked to the interoceptive awareness and which is the patient's ability to relax through the measurement of the hearth rate variability (HRV).

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic nonspecific low back pain for at least three months
* Subjects aged between 18 and 50 years

Exclusion Criteria:

* Presence of acute low back pain
* Low back pain due to other causes (vertebral fractures, spondylolisthesis, herniated discs, lumbar canal stenosis)
* Disorders of central and/or peripheral nervous system
* Systemic inflammatory disease (eg rheumatoid arthritis)
* Systemic infectious disease
* Neoplastic disease
* Previous Surgery
* Cognitive impairment
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change of Visual Analogue Scale (VAS) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It is a scale for the assessment of pain and it's based on a ten point scale, where 0 means no pain and 10 the greatest pain ever both at rest and during movements.

SECONDARY OUTCOMES:
Change of McGill Pain Questionnaire from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  This scales evaluates the degree of functional impairment in activities of daily life caused by pain. It consist of ten sections including pain intensity, personal care, lifting, walking, sitting standing, sleeping, sex, social life and travelling. Each section includes six sentences relating to different level of limitation in the same activity (0: no limitation, 5: maximal limitation).
Change of Multidimensional Assessment of Interoceptive Awareness (MAIA) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  The questionnaire is divided into 32 items organized into eight subcategories consisting of three to seven items each. The subcategories measure: the awareness of unpleasant, pleasant or neutral body sensations, the tendency not to ignore the feelings of pain or discomfort, not to worry about painful sensations or discomfort, the ability not to draw attention away from body sensations, awareness of the existence of connections between body sensations and emotional status, the ability to control the psychological stress by focusing on body sensations, the ability to listen to your body and the belief that the experiences coming from your body are safe and reliable. It 'a multidimensional assessment questionnaire and self-administered. For each subcategory, the patient may express a score from 0 (never) to 5 (always), the highest score corresponds to a higher level of awareness.
Change of SF-12 Health Survey Questionnaire from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  The questionnaire consist in twelve questions that explore eight sub-categories that measure the physical activity, role limitations due to physical health and emotional state, physical pain, the perception of general health, vitality, social activities, mental health and changes in health status and two indices that summarize the overall assessment of the subject with respect to his physical health (ISF) and mental (ISM).
Change of Waddell Disability Index from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It includes nine parameters: pain experienced in a sitting position, travelling, standing,walking and lifting weights and the need to put on or remove footwear, sleep disturbance, life restriction and sex life restriction to measure. The maximum score is 9 points. A score > 5 indicates significant disability.
Change of hearth rate variability (HRV) expressed as coherent ratio from baseline to 4 weeks | baseline, 4 weeks
  Its an index monitored by a plethysmograph that records the heart rate variability (variation in the time interval between a heartbeat and the other) a parameter capable of expressing a person's level of stress through the coherence ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Maria Saraceni, Principal Investigator — Umberto I Hospital, University "Sapienza" of Rome
Locations (1):
- Umberto I Hospital, Rome, Italy